CLINICAL TRIAL: NCT05214118
Title: Project BETTER: Bringing Education Through Technology, Empathic Listening, and Research - A Feasibility Randomized Controlled Trial
Brief Title: Bringing Education Through Technology, Empathic Listening, and Research
Acronym: BETTER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HM20023314
Record Dates: First submitted 2022-01-10; First posted 2022-01-28 (Actual); Results first posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-06

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brochure (No Intervention)
- Technology-based program (Experimental)
  Interventions: Behavioral: technology-based program

INTERVENTIONS:
Behavioral: technology-based program — Participants will be asked to complete three 25-minute modules covering the transition from pregnancy to postpartum, possible neonatal abstinence syndrome (NAS) or neonatal withdrawal syndrome (NOWS), and interactions with child welfare.
  Arms: Technology-based program

SUMMARY:
The purpose of this study is to test a new educational technology-based program and brochure as a supplement to prenatal education from providers. The program provides education about common challenges that pregnant and parenting women receiving medication for Opioid Use Disorder (OUD) often face. Specifically, it addresses the transition from pregnancy to postpartum, possible neonatal abstinence syndrome (NAS) or neonatal withdrawal syndrome (NOWS), and interactions with child welfare.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. ≥18 years of age
3. Meet criteria for Opioid Use Disorder
4. Currently receiving MOUD pharmacotherapy (including buprenorphine, buprenorphine/naloxone, or methadone)
5. Pregnant (<34 weeks EGA)
6. Initial in-person visit at OB MOTIVATE clinic for the current pregnancy ≤10 weeks ago

Exclusion Criteria:

1. Considering/planning adoption
2. Present with a serious cognitive/psychiatric impairment
3. Existing language barriers making true informed consent impossible

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant females
Enrollment: 29 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin E Martin, MD, MPH, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Brochure: No intervention, brochure
Period: Overall Study
Arm/Group | Brochure | Technology-based Program
Started | 13 | 16
Completed | 11 | 13
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 0 | 2
Not completed — delivered late preterm 34 wks gestation | 1 | 1
Not completed — moved | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brochure | Technology-based Program | Total
Number analyzed (Participants) | 13 | 16 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 16 | 29
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.3 (5.3) | 29.7 (3.6) | 30 (4.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 29
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 12 | 16 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 6 | 9
  White | 10 | 9 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 16 | 29

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of the Intervention
Description: Participants will complete a survey about the feasibility of the intervention consisting of 4 items rated on a 0 to 6 scale. Scores will be summed to yield a final feasibility score ranging from 0 to 24. Higher scores indicate higher feasibility.
Time Frame: Within 2 weeks of completing the intervention
Population: Participants will complete a survey about the feasibility of the intervention consisting of 4 items rated on a 0 to 6 scale. Scores will be summed to yield a final feasibility score ranging from 0 to 24. Higher scores indicate higher feasibility.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brochure | Technology-based Program
Number analyzed (Participants) | 11 | 13
score on a scale | 21.5 (2.3) | 21.2 (2.9)

2. Primary Outcome: Acceptability of the Intervention
Description: Participants will complete a survey about the acceptability of the intervention consisting of 10 items rated on a 1 to 5 scale. Higher scores indicated higher acceptability.
Time Frame: Within 2 weeks of completing the intervention
Population: Participants will complete a survey about the acceptability of the intervention consisting of 10 items rated on a 1 to 5 scale. Scores will be summed to yield a final feasibility score ranging from 10 to 50. Higher scores indicated higher acceptability.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brochure | Technology-based Program
Number analyzed (Participants) | 11 | 13
score on a scale | 47.6 (5.5) | 48.3 (7.6)

3. Secondary Outcome: Change in Perceived Competence
Description: Participants will complete a survey assessing their feelings of competence related to the information covered by the intervention. The items will be rated on a 1 to 7 scale. Higher scores indicated higher perceived competence. An increase in perceived competence suggests a greater sense of confidence, mastery, and belief in one's ability to achieve goals within that area. This can be linked to positive outcomes like improved performance, motivation, and goal attainment. A decrease in perceived competence indicates a diminished sense of self-efficacy and belief in one's abilities, potentially leading to reduced motivation, avoidance of challenges, and lower engagement.
Time Frame: Baseline to within 2 weeks of completing the intervention, up to 5 weeks
Population: Participants will complete 12 items (4 items per 3 content areas) assessing their feelings of competence related to the information covered by the intervention. The items will be rated on a 1 to 7 scale. Higher scores indicated higher perceived competence.
Measure: Mean (Standard Deviation); unit: mean score on a scale
Arm/Group | Brochure | Technology-based Program
Number analyzed (Participants) | 12 | 9
mean score on a scale | .75 (9.7) | .3 (8.5)

4. Secondary Outcome: Change in Parental Competence
Description: Participants will complete a survey assessing their feelings of competence related to the parenting. The items will be rated on a 1 to 6 scale. An increase in perceived competence suggests a greater sense of confidence, mastery, and belief in one's ability to achieve goals within that area. This can be linked to positive outcomes like improved performance, motivation, and goal attainment. A decrease in perceived competence indicates a diminished sense of self-efficacy and belief in one's abilities, potentially leading to reduced motivation, avoidance of challenges, and lower engagement.
Time Frame: Baseline to within 2 weeks of completing the intervention, up to 5 weeks
Population: Participants will complete a 16-item survey assessing their feelings of competence related to the parenting. The items will be rated on a 1 to 6 scale. Higher scores indicated higher perceived parental competence.
Measure: Mean (Standard Deviation); unit: mean score on a scale
Arm/Group | Brochure | Technology-based Program
Number analyzed (Participants) | 12 | 10
mean score on a scale | 3.3 (9) | -1.5 (11.5)

ADVERSE EVENTS:
Time Frame: February 2022-October 2023 overall for the study. During the duration of study involvement individually for each subject which is Baseline to within 2 weeks of completing the intervention, up to 5 weeks.
Arm/Group | Brochure | Technology-based Program
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/16
Serious Adverse Events (participants affected / at risk) | 1/13 | 0/16
Other Adverse Events (participants affected / at risk) | 0/13 | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brochure (N=13) | Technology-based Program (N=16)
Cardiac disorders (Cardiac disorders) | 1 (1) | 0 (0) — Participant was placed on extracorporeal membrane oxygenation and had to be ventilated, participants fetus did not survive.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT05214118/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-07): https://cdn.clinicaltrials.gov/large-docs/18/NCT05214118/ICF_001.pdf